CLINICAL TRIAL: NCT07077109
Title: Continuous Non-invasive Electrophysiological Monitoring During Maternal Exercise: a Feasibility Study
Brief Title: Feasibility Study: Continuous Fetal Monitoring During Maternal Exercise
Acronym: NIEM-S
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Phebe Berben, Medical doctor, PhD Candidate, Coordinating Investigator NIEM-S study, Maxima Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL009785
Record Dates: First submitted 2025-04-22; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Monitoring
Keywords: Electrophysiological monitoring; Pregnancy; Sport; Feasibility study; Maternal exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrophysiological monitoring (Experimental): See intervention
  Interventions: Device: Electrophysiological monitoring

INTERVENTIONS:
Device: Electrophysiological monitoring — electrofysiological CTG monitoring with the Nemo Fetal Monitoring System (Nemo Healthcare B.V., Veldhoven, the Netherlands). The NFMS consists of a wireless and beltless electrode patch on the maternal abdomen. It monitors fetal heart rate by fetal electrocardiography, maternal heart rate by maternal electrocardiography and the electrical activity of the uterine muscle by electrohysterography.

SUMMARY:
This feasibility study will be the first study to assess the feasibility of continuous electrophysiological monitoring during maternal exercise in women with an uncomplicated pregnancy. This may help to better understand fetal condition during exercise and offer personalised exercise recommendations in the future. In future, validating the feasibility and safety of exercise could promote greater exercise engagement among pregnant women and increase fetal wellbeiing.

DETAILED DESCRIPTION:
The Nemo Fetal Monitoring Sytem (Nemo Healthcare B.V., Veldhoven, the Netherlands) will be used for electrophysiological monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years old
* Pregnant women with an uncomplicated singleton pregnancy and a gestational age between 30+0 and 40+0 weeks and days
* Oral and written informed consent is obtained
* Engage in aerobic exercise during pregnancy

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Insufficient knowledge of Dutch or English language
* Women with a multiple pregnancy
* Contra-indications for the Nemo Fetal Monitoring System (NFMS):

  * Fetal and/or maternal cardiac arrhythmias
  * Contraindications to abdominal placement (dermatologic diseases of the abdomen precluding preparation of the abdomen with abrasive paper)
  * Women connected to an external or implanted electrical stimulator, such as a pacemaker (because of disturbance of the electrophysiological signal)
* Fetus with known congenital or chromosomal abnormalities
* Women with absolute or relative contraindications to aerobic exercise during pregnancy at time of inclusions and during maternal exercise:

  * Mild or severe respiratory diseases (e.g. chronic obstructive pulmonary disease, restrictive lung disease and cystic fibrosis)
  * Mild or severe acquired or congenital heart disease with exercise intolerance
  * Uncontrolled or severe arrhythmia
  * Vasa previa
  * Type 1 diabetes
  * IUGR
  * Severe PE
  * Cervical insufficiency
* Women with relative contraindications to aerobic exercise during pregnancy:

  * Mild respiratory disorders
  * Mild congenital or acquired heart disease
  * Well-controlled type 1 diabetes
  * Pre-eclampsia
  * Cervical insufficiency
  * Placenta previa
  * Untreated thyroid disease
  * Symptomatic, severe eating disorder
  * Multiple nutrient deficiencies and/or chronic undernutrition
  * Moderate-heavy smoking (> 20 cigarettes per day)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Success rate of continuous electrophysiolgoical monitoring during maternal exercise | 15 minutes (min) before, 30 min during and 15 min after maternal exercise
  Defined as the percentage of time during continuous maternal exercise with concurrent signal output of the fetal heart rate. Continous electrophysiological monitoring is feasible by a successrate of =>80%

SECONDARY OUTCOMES:
Maternal heartrate | 15 min before, 30 min during and 15 min after maternal exercise
  Mean maternal heart rate in beats per minutes (bpm) from cardiotocogram
Mean maternal heartrate | 15 min before, 30 min during and 15 min after maternal exercise
  Mean maternal heart rate in bpm from cardiotocographic output
Fetal heart rate variability | 15 min before, 30 min during, 15 min after exercise
  Fetal heart rate variability from cardiotocogram, measured as average short term variability and average long term variability
Fetal heart rate | 15 min before, 30 min during and 15 min after maternal exercise
  Mean fetal heart rate in bpm from cardiotocogram
Contraction frequency | 15 min before, 30 min during and 15 min after maternal exercise
  Mean contraction freqency from cardiotocogram, defined as the number of contractions per 10 minutes.
Contraction duration | 15 min before, 30 min during and 15 min after maternal exercise
  Mean contraction duration in seconds from cardiotocogram
Contraction intensity | 15 min before, 30 min during and 15 min after maternal exercise
  Mean maximum contraction intensity (i.e. amplitude) from cardiotocogram (in arbitrary units)
Contraction interval | 15 min before, 30 min during and 15 min after maternal exercise
  Mean contraction interval in seconds, from cardiotocogram
Accelerations | 15 min before, 30 min during and 15 min after maternal exercise
  Increase in the fetal heart rate above the baseline lasting 10-120 seconds and reaching a peak of at least 10 seconds, from cardiotocogram
Decelerations | 15 min before, 30 min during and 15 min after maternal exercise
  Decrease in fetal heart rate under the baseline lasting at 15 seconds, and with a minimum amplitude of 15 seconds, from cardiotocogram.
Signal loss | 15 min before, 30 min during and 15 min after maternal exercise
  Percentage of fetal heart rate signals values under 35bpm, from cardiotocogram
Maternal satisfaction of continuous fetal monitoring and tolerability of the patch during exercise | Directly after exercise (duration to complete: 10 min)
  Maternal satisfaction by selfmade questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Simone Goossens, PhD, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication